CLINICAL TRIAL: NCT00914758
Title: Comparison of Alemtuzumab (Campath®) and High Dose Interferon Beta-1a (Rebif®) Treatment on Cognition in Subjects With Relapsing Forms of MS
Brief Title: Comparison of Campath and Rebif Treatment on Cognition in Multiple Sclerosis (MS)
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Washington Neuropsychology Research Group (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Jeffrey Wilken, Ph.D./Executive Director, Washington Neuropsychology Research Group
Other Study IDs: WNRG02
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Last update posted 2009-06-05 (Estimated); Status verified 2009-06

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: multiple sclerosis; cognition; cognitive functioning; Campath; Rebif; alemtuzumab; interferon
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- MS patients on Campath®: This group is comprised of patients diagnosed with relapsing remitting multiple sclerosis who were assigned to the Campath® treatment arm of the Care-MS II trial, for which this study is a sub-study
- MS patients on Rebif®: This group is comprised of patients diagnosed with relapsing remitting multiple sclerosis who were assigned to the Rebif® treatment arm of the Care-MS II trial, for which this study is a sub-study
- Control group: This group is comprised of non-MS, non-CNS compromised control participants matched in age, education level, and socioeconomic status to the participants in the 2 MS treatment groups

SUMMARY:
People with multiple sclerosis (MS) often experience problems with cognitive functioning, which can be debilitating and interfere with their daily functioning. However, research has shown that MS disease modifying agents have had some success in treating cognitive problems. The main purpose of this research study is to investigate how well two medicines (alemtuzumab (Campath®) and interferon beta-1a (Rebif®)) work in treating MS-related cognitive problems (e.g., attention, memory, speed of thinking). Participants enrolled will be assessed prior to their first study-related medication dose and re-assessed throughout treatment. It is expected that participants taking Campath® will demonstrate relative stability in cognitive functioning relative to those taking Rebif®. Specifically, the cognitive performance of Rebif® participants will decline somewhat over time, but the cognitive performance of Campath® participants will remain stable.

DETAILED DESCRIPTION:
The current will use a neuropsychological evaluation capable of detecting the broad range of cognitive difficulties associated with relapsing remitting MS (RRMS). It is a sub-study of an investigation already underway, called Care-MS II, in which participants diagnosed with RRMS are treated with either Campath® or Rebif®. We will observe those participants already assigned to one of the two study arms in Care-MS II and compare cognitive functioning over time of those taking Campath® and those taking Rebif®. We will also compare the change in cognitive functioning for each active group to that of a matched control group. This will help to control for practice effects and help to establish whether either medication helps to truly stabilize cognitive decline (i.e., relative to non-MS controls). We will obtain neurocognitive data at baseline (prior to the first study dose of Campath® or Rebif®), 12 months (before second dose for Campath® participants), 14 months (2 months after the second dose for Campath® participants), 24 months (prior to the third dose for Campath® participants), and 26 months (2 months after the third dose for Campath® participants). The neurocognitive battery will include gold-standard traditional neuropsychology measures as well as newer, validated computerized measures capable of detecting changes in attention and processing speed that are often missed by traditional measures. Since participants in Care-MS II will also have MRI data at baseline, 1 year, and 2 years, cognitive findings will be correlated with MRI data and analyzed in a post-hoc, exploratory manner for the participants with MS.

Hypotheses include:

* 1: Participants taking Campath® will demonstrate relative stability in cognitive functioning relative to those taking Rebif®. Specifically, the cognitive performance of Rebif® participants will decline somewhat over time, but the cognitive performance of Campath® participants will remain stable.
* 2: Participants taking Campath® will demonstrate similar cognitive change (i.e., change in scores over 2 years) as normal, matched controls.
* 3: Participants taking Rebif® will demonstrate greater cognitive change (i.e., change in scores over 2 years) as compared to normal, matched controls.
* 4: Cognitive stability in Campath® participants will correlate with stability in MRI parameters.
* 5: Cognitive change in Rebif® participants will correlate with greater activity on MRI parameters.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing remitting MS and enrollment in Care-MS II trial
* Non-MS controls must be neurologically healthy (with respect to conditions that impact CNS functioning).
* Participants must be between the ages of 25 and 50.
* Corrected vision of subjects must be no worse than 20/50.
* Participants must have at least 10 years of education.
* Participants must be capable of writing and pressing the buttons on a computer mouse.
* Participants must be capable of understanding and following all test instructions.

Exclusion Criteria:

* Participants with a history of head injury, seizures, or neurological conditions involving the central nervous system (other than MS for the MS groups).
* Participants with upper extremity dysfunction which prohibits them from using a computer mouse.
* Participants who are colorblind.
* Participants with history of psychosis or other severe mental illness.
* Participants with current alcohol/substance abuse.
* Participants taking medications with potential adverse CNS effects

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: community sample diagnosed with relapsing remitting multiple sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2009-03; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Paced Auditory Serial Addition Test | Prior to first study-related medication dose and re-assessed at 12 months, 14 months, 24 months, and 26 months
Stroop Test | Prior to first study-related medication dose and re-assessed at 12 months, 14 months, 24 months, and 26 months
Symbol Digit Modalities Test | Prior to first study-related medication dose and re-assessed at 12 months, 14 months, 24 months, and 26 months
Lexical and Categorical Associative Fluency Tests | Prior to first study-related medication dose and re-assessed at 12 months, 14 months, 24 months, and 26 months
Automated Neuropsychological Assessment Metrics | Prior to first study-related medication dose and re-assessed at 12 months, 14 months, 24 months, and 26 months
MS Quality of Life Instrument-54 | Prior to first study-related medication dose and re-assessed at 12 months, 14 months, 24 months, and 26 months
Fatigue Severity Scale | Prior to first study-related medication dose and re-assessed at 12 months, 14 months, 24 months, and 26 months
Epworth Sleepiness Scale | Prior to first study-related medication dose and re-assessed at 12 months, 14 months, 24 months, and 26 months
MS Fatigue Impact Scale | Prior to first study-related medication dose and re-assessed at 12 months, 14 months, 24 months, and 26 months

SECONDARY OUTCOMES:
MRI data | prior to first study-related medication dose and reassessed at 1 year and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Wilken, Ph.D., Principal Investigator — Washington Neuropsychology Research Group
Locations (7):
- United States (7):
  - The Research and Education Institute of Alta Bates Summit Medical Center, Berkely, California
  - Associates In Neurology. PSC, Lexington, Kentucky
  - Springfield Neurology Associates, LLC, Springfield, Massachusetts
  - Dartmouth Medical School/Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Multiple Sclerosis Center of NE New York, Empire Neurology, PC, Latham, New York
  - Multiple Sclerosis Center, University of Rochester Medical Center, Rochester, New York
  - MS Center of Greater Washington, Vienna, Virginia